CLINICAL TRIAL: NCT06601881
Title: Investigation of the Effects of Thorocal Mobilization and Diaphragmatic Breathing Training on Postural Stability and Target Consistency in Archery.
Brief Title: The Effects of Thoracic Mobilization and Diaphragmatic Breathing on Postural Sway in Archers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Sağlık ve Teknoloji Üniversitesi (Other)
Responsible Party: Principal Investigator, Gamze Aydoğan, Lecturer, Kocaeli Sağlık ve Teknoloji Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 09.23.1196
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: PERFORMANCE-ENHANCING EFFECT
Keywords: ARCHERY; postural stability; diaphragmatic breathing training; thoracal mobilization exercises
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group- Group I (Experimental): individuals will do thoracic mobilization exercises and Diaphragmatic Breathing Training
  Interventions: Other: Experimental
- Control group- Group II (Active Comparator): Control Group will do plasebo Diaphragmatic Breathing Training and plaseboThoracic mobilization exercises
  Interventions: Other: Control (placebo) group

INTERVENTIONS:
Other: Experimental — Thoracic mobilization exercises will include:
  1. Thoracic Spine Extension exersice
  2. Thoracic rotation exersice
  3. Cat-Camel Exercise
  4. Lateral Flexion of the Thoracic Spine
  5. Muscules Psoas Stretching
  6. Diaphragm Release Technique
  Diaphragmatic Breathing Training will include:
  1. Diaphragmatic Breathing
  2. Crocodile Breathing Technique
  3. Breathing with an exercise band
  4. Pursed lip breathing
  Other Names: Thoracic mobilization exercises and Diaphragmatic Breathing Training
  Arms: Experimental Group- Group I
Other: Control (placebo) group — Placebo Thoracic mobilization exercises will include:
  1. Placebo Thoracic Spine Extension exersice
  2. Placebo Thoracic rotation exersice
  3. Placebo Cat-Camel Exercise
  4. Placebo Lateral Flexion of the Thoracic Spine
  5. Placebo Muscules Psoas Stretching
  6. Placebo Diaphragm Release Technique
  Placebo Diaphragmatic Breathing Training will include:
  1. Placebo Diaphragmatic Breathing
  2. Placebo Crocodile Breathing Technique
  3. Placebo Breathing with an exercise band
  4. Placebo Pursed lip breathing
  Arms: Control group- Group II

SUMMARY:
Shooting in archery requires tremendous postural stability to minimize oscillations when the upper body area is under high muscle tension. Postural oscillations depend especially on the alignment of the target and the arrow and the center of gravity being within the base of support. In addition, it has been reported that heart rate changes and breathing patterns affect postural control and therefore performance. Increasing pulse values during shooting negatively affect shooting performance by causing increased postural oscillations and body shaking. The breathing pattern directly affects postural oscillations by affecting the heart rate.It has been reported that the diaphragm has important effects on breathing and trunk control due to its anatomical connections and that the diaphragm movement during breathing is synchronized with the stabilization function. During breathing, the diaphragm descends into the abdominal cavity, causing a positive pressure increase in the intra-abdominal region. Due to this increasing pressure, it expands the abdominal area to the limit allowed by the abdominal muscles and the abdominal wall. Then, with the eccentric contraction of the abdominal muscles, the descent of the diaphragm is blocked at a certain point and the abdominal muscles resist the movement of the diaphragm. In response to this counter-reaction, the diaphragm realizes inspiration by providing a 3-dimensional expansion by opening the lower ribs to the posterolateral. It has been reported that the stabilization effect of the diaphragm is the result of its contraction especially towards these sides, therefore a good level of thoracic mobilization will increase the lateral contraction capacity of the diaphragm. This is ultimately associated with a stronger stabilization effect. On the other hand, impairment of synchronization may result in spinal segments being under excessive stress and reducing stability. Studies in patients and healthy individuals have shown that diaphragmatic breathing contributes to balance by increasing the strength of the diaphragm and deep core muscles. Shooting performance in archery is closely related to the correct breathing pattern and diaphragmatic movement, as it is affected by trunk mobility and postural stability. On the other hand, when we look at the contents of archery training, there are general condition-increasing exercises, special muscle strengthening exercises, methods for developing mental skills and techniques, and methods such as diving and bungee jumping as new training methods. It was observed that exercises were not included in the training programs. The aim of this study is to investigate the scope of postural stability and target stability of thoracic mobilization techniques and diaphragmatic breathing training in order to reveal the stabilization level of the diaphragm at the optimum level in archers.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* Individuals over the age of 18
* Individuals have been practicing archery for at least 2 years and
* Individuals have a WA (World Archery Federation) score between 360-570

Exclusion Criteria:

* Surgery in the trunk, upper extremities, neck and lower back within the last 1 year,
* Athletes who have sustained injuries to the trunk, upper limbs, lower back and neck in the last 6 months,
* Athletes who have suffered from respiratory system diseases such as pneumonia, acute bronchitis, etc. that may affect respiratory capacity within the last 1 year
* Athletes with chronic respiratory system diseases (asthma, emphysema, chronic bronchitis, etc.) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
measurement of anterior-posterior, medio-lateral sway | will be measured at initially,6 week and 10 week
  The data obtained with the force platform will be analyzed using Matscan 7.10 software and the center of gravity movement area - COF area/cm²; Anteroposterior sway/cm; Side sway-mediolateral sway/cm values, center of pressure displacement rate-VCP, mm/s-statokinesiogram area-mm² will be determined.
measurement of total score from archers shots | will be measured at ınitially, 6 week and 10 week
  As a result of shooting 60 arrows on the target board, the points will be added up and the total score will be obtained.

SECONDARY OUTCOMES:
measurement of Maximum inspiratory pressure (MİP-MEP) | changes of Maximum inspiratory pressure( Maximum inspiratory pressure and Maximum expiratory pressure) will be measured at ınitially, 6 week and 10 week
  maximum inspiratory pressure and maximum expiratory pressure will be mesured by MicroRPM device

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Aydoğan, MsC, PT, Principal Investigator — PhD student; Nilüfer Kablan, asst. Prof, Principal Investigator — head of physical medicine and rehabilitation department; Yaşar Tatar, Prof. MD, Study Director — Professor at the Faculty of Sports Sciences